CLINICAL TRIAL: NCT06758700
Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of Teniposide as a Post-Line Therapy for c-Myc-Driven Extensive-Stage Small Cell Lung Cancer
Brief Title: Post-line Treatment With Teniposide for c-Myc-driven Extensive-stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Collaborators: CHINA RESOURCES DOUBLE-CRANE PHARMACEUTICAL CO.,LTD (Unknown)
Responsible Party: Principal Investigator, Ren Shengxiang, Prof., Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VM26-201; ChiCTR2400094090 (Other: Chinese Clinical Trial Registry)
Record Dates: First submitted 2024-12-26; First posted 2025-01-06 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC); Thoracic Neoplasms; Lung Neoplasms; Lung Diseases
Keywords: c-Myc; SCLC; Phase II; Post-line
MeSH Terms: conditions — Small Cell Lung Carcinoma; Thoracic Neoplasms; Lung Neoplasms; Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teniposide group (Other): Teniposide administration
  Interventions: Drug: Teniposide administration

INTERVENTIONS:
Drug: Teniposide administration — Teniposide administration: 60mg/m2, diluted with 500ml of 0.9% sodium chloride injection before use, intravenous infusion for more than 1 hour, for 3-5 consecutive days, with 21 days as one cycle of treatment.

SUMMARY:
The study is being conducted to investigate the efficacy and safety of teniposide in patients with extensive-stage small cell lung cancer who have failed standard treatment and with high expression of the c-Myc-driven FBXW2/MYC gene. Based on the results, the study will explore the correlation between the expression of FBXW2/MYC and the efficacy of teniposide.

ELIGIBILITY:
Inclusion Criteria:

1. extensive stage small cell lung cancer
2. Progression after receiving at least one chemotherapy drug treatment in the past;
3. ECOG score 0-1
4. c-Myc-driven
5. Expected survival period ≥3 months
6. Age: 18-75 years old;
7. The informed consent form complies with the ICH-GCP principles.

Exclusion Criteria:

1. No measurable lesions
2. Other severe and persistent diseases or organ system dysfunction;
3. Women planning pregnancy or men planning family planning;
4. Women who are pregnant or breastfeeding;
5. Those who cannot follow the research protocol provided by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Image evaluations were conducted at baseline and every 6-8 weeks after the administration of teniposide, through study completion, an average of 1 year

SECONDARY OUTCOMES:
Disease Control Rate | Image evaluations were conducted at baseline and every 6-8 weeks after the administration of teniposide, through study completion, an average of 1 year
Progression Free Survial | Image evaluations were conducted at baseline and every 6-8 weeks after the administration of teniposide, until progression or death, an average of 1 year
Duration of Response | Image evaluations were conducted at baseline and every 6-8 weeks after the administration of teniposide, until progression or death, an average of 1 year
Adverse events(AEs), serious adverse events（SAEs）as assessed by CTCAE v5.0 | From Baseline up to 30 days after the last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Postmus PE, Haaxma-Reiche H, Smit EF, Groen HJ, Karnicka H, Lewinski T, van Meerbeeck J, Clerico M, Gregor A, Curran D, Sahmoud T, Kirkpatrick A, Giaccone G. Treatment of brain metastases of small-cell lung cancer: comparing teniposide and teniposide with whole-brain radiotherapy--a phase III study of the European Organization for the Research and Treatment of Cancer Lung Cancer Cooperative Group. J Clin Oncol. 2000 Oct 1;18(19):3400-8. doi: 10.1200/JCO.2000.18.19.3400. PMID 11013281
- [Background] Postmus PE, Smit EF, Haaxma-Reiche H, van Zandwijk N, Ardizzoni A, Quoix E, Kirkpatrick A, Sahmoud T, Giaccone G. Teniposide for brain metastases of small-cell lung cancer: a phase II study. European Organization for Research and Treatment of Cancer Lung Cancer Cooperative Group. J Clin Oncol. 1995 Mar;13(3):660-5. doi: 10.1200/JCO.1995.13.3.660. PMID 7884426
- [Background] Liu Q, Zhang J, Guo C, Wang M, Wang C, Yan Y, Sun L, Wang D, Zhang L, Yu H, Hou L, Wu C, Zhu Y, Jiang G, Zhu H, Zhou Y, Fang S, Zhang T, Hu L, Li J, Liu Y, Zhang H, Zhang B, Ding L, Robles AI, Rodriguez H, Gao D, Ji H, Zhou H, Zhang P. Proteogenomic characterization of small cell lung cancer identifies biological insights and subtype-specific therapeutic strategies. Cell. 2024 Jan 4;187(1):184-203.e28. doi: 10.1016/j.cell.2023.12.004. PMID 38181741
- [Background] Dhanasekaran R, Deutzmann A, Mahauad-Fernandez WD, Hansen AS, Gouw AM, Felsher DW. The MYC oncogene - the grand orchestrator of cancer growth and immune evasion. Nat Rev Clin Oncol. 2022 Jan;19(1):23-36. doi: 10.1038/s41571-021-00549-2. Epub 2021 Sep 10. PMID 34508258
- [Background] Sabari JK, Lok BH, Laird JH, Poirier JT, Rudin CM. Unravelling the biology of SCLC: implications for therapy. Nat Rev Clin Oncol. 2017 Sep;14(9):549-561. doi: 10.1038/nrclinonc.2017.71. Epub 2017 May 23. PMID 28534531
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338